CLINICAL TRIAL: NCT00138099
Title: Dalteparin's Influence on Renally Compromised: Anti-Ten-A Study (DIRECT)
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Critical Care Trials Group (Other); Pfizer (Industry)
Organization: McMaster University (Other)
Other Study IDs: 092103; File No: 9427-M1133-21C; Control No: 092103
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2006-11

CONDITIONS: Renal Insufficiency
Keywords: Critically ill patients (ICU); Deep Venous Thromboembolism prevention; Renal Failure; Critically ill
MeSH Terms: conditions — Renal Insufficiency; Critical Illness | interventions — Dalteparin

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fragmin (dalteparin sodium)

SUMMARY:
The investigators' primary research objective is:

* To determine the safety of dalteparin prophylaxis, 5,000 IU once-daily, in Intensive Care Unit (ICU) patients based on:

  * the proportion of patients with trough anti-Xa > 0.40 IU/mL during dalteparin prophylaxis after 3 + 1 days, 10 + 1 days, and 17 + 1 days of dalteparin prophylaxis;
  * the risk of major bleeding during the treatment period.

The investigators' secondary research objectives are:

* To determine the pharmacokinetic properties of dalteparin prophylaxis in ICU patients with severe renal insufficiency;
* To identify clinical and laboratory factors that predict an excessive anticoagulant effect (anti-Xa > 0.10 IU/mL);
* To estimate the relationship between trough anti-Xa levels and bleeding.

The DIRECT Pilot Study:

Before embarking on a large trial of low molecular weight heparin (LMWH) versus standard unfractionated heparin (UFH), the DIRECT Study is needed to observe whether bioaccumulation of LMWH occurs in ICU patients with moderate to severe renal insufficiency, and to address potential problems with protocol implementation.

DETAILED DESCRIPTION:
Critically ill patients who are admitted to an intensive care unit (ICU) are at high risk for deep vein thrombosis (DVT), with an estimated 20-40% of patients developing DVT without prophylaxis. Preventing DVT is important because DVT is usually clinically silent in such patients, and its first manifestation may be life-threatening pulmonary embolism.

About 30% of ICU patients have renal insufficiency, based on a calculated creatinine clearance (CrCl), and such patients have 4-fold higher risk of DVT than those with normal renal function.

The current anticoagulant regimen that is used to prevent DVT in such patients, consisting of unfractionated heparin (UFH), 5000 IU twice-daily, may be inadequate.

A recent prospective cohort study by our research group that investigated the risk of DVT in 261 ICU patients found that 10% of patients developed proximal vein DVT after admission to the ICU despite receiving UFH, 5000 IU twice-daily.

In other patient groups at high risk for DVT, low-molecular-weight heparins (LMWHs) have replaced UFH for DVT prophylaxis because of superior efficacy.

Despite superior efficacy and safety in many patients, there is concern about using LMWHs in patients with renal insufficiency because LMWHs are cleared by the kidney. LMWH use in such patients might result in an excessive anticoagulant effect, with the potential to increase bleeding.

Much of the concern about the safety of LMWH in patients with renal insufficiency pertains to therapeutic-dose LMWH used to treat DVT. Prophylactic-(or low) dose LMWH that is used to prevent DVT in ICU patients is about 25-33% of a therapeutic-dose.

Three sources of evidence suggest that prophylactic-dose LMWH may be safe in patients with renal insufficiency. First, current evidence does not support the fact that prophylactic-dose LMWH accumulates and should be avoided in such patients. Second, prophylactic-dose LMWH appears to be safe in hemodialysis patients. Third, preliminary work by our research group suggests that dalteparin, 5000 IU once-daily, does not accumulate in ICU patients with renal insufficiency. Thus, 0 of 10 ICU patients with a CrCl <50 mL/min/1.73m2 who received dalteparin had a detectable trough anticoagulant effect (anti-Xa >0.10 IU/mL). Further, when the relationship between CrCl and peak anti-Xa levels was assessed, there was no correlation (r<0.2). Finally, in 2 patients with severe renal insufficiency (CrCl<30 mL/min/1.73m2) who received dalteparin, 5000 IU once-daily, all 9 trough anti-Xa values were <0.10 IU/mL.

No study has investigated the safety of low-dose LMWH in ICU patients with impaired renal function; until such a study is completed, randomized trials assessing the efficacy of low-dose LMWH for DVT prophylaxis among ICU patients will not be feasible.

As a first step in addressing this problem, we propose an open-label pilot study to assess the safety of dalteparin prophylaxis, 5000 IU once-daily, in ICU patients with severe renal insufficiency.

The safety of the proposed dalteparin prophylaxis regimen will be assessed by determining the risk of an excessive anticoagulant effect and the risk of major bleeding. Dalteparin prophylaxis will be considered safe if 2 criteria are satisfied by the end of the treatment period:

* proportion of patients with trough anti-Xa level >0.40 IU/mL is ~10% or less (exclude 17% with 95% confidence);
* risk of major bleeding is ~4% or less (exclude 10% with 95% confidence).

If we show that dalteparin prophylaxis is safe in ICU patients with severe renal insufficiency, this will improve patient care in 2 ways:

* dalteparin may reduce the risk of DVT (although this should be tested in future trials); and
* dalteparin would reduce heparin induced thrombocytopenia (HIT), an infrequent but serious complication of UFH.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged > 18 years
* Admitted to an ICU with an expected ICU length of stay > 72 hours
* Severe renal insufficiency, defined by a calculated CrCl < 30 mL/min/1.73m2

Exclusion Criteria:

* ICU admission for > 2 weeks at time of screening
* ICU admission within 3 months of cardiac surgery or neurosurgery
* Active bleeding or at high risk for bleeding complications
* Thrombocytopenia (platelet count < 75 x 10^9/L) at time of screening
* Coagulopathy (International Normalized Ratio [INR] or activated partial thromboplastin time [aPTT] > 2 times upper limit of normal) at time of screening
* Patient had an indwelling epidural catheter for epidural analgesia within the last 12 hours
* Receipt of > 2 doses of LMWH (prophylactic- or therapeutic-dose) in the ICU
* Receiving or requiring therapeutic-dose anticoagulation (eg., deep vein thrombosis [DVT]) at time of screening
* Receiving dialysis that requires anticoagulation (eg., PRISMA, slow continuous ultrafiltration [SCUF]) at time of screening
* Weight < 45 kg
* Woman who is pregnant or lactating
* Bilateral lower limb amputation
* Previous adverse reaction to heparin or LMWH (eg., allergy, heparin-induced thrombocytopenia [HIT])
* Contraindication to receiving blood products
* Life expectancy < 14 days or receiving palliative care
* Prior enrolment in this study or enrolment in a concurrent related clinical trial
* Patient or surrogate decision-maker does not provide consent to participate in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2004-07; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Douketis, MD, Principal Investigator — McMaster University; Deborah J Cook, MD, Principal Investigator — McMaster University
Locations (14):
- Canada (14):
  - Queen Elizabeth II Health Science Centre, Halifax, Nova Scotia
  - Hamilton Health Science Centre - Hamilton General Hospital, Hamilton, Ontario
  - Hamilton Health Science Centre - McMaster University, Hamilton, Ontario
  - St Joseph's HealthCare, Hamilton, Ontario
  - Hamilton Health Science Centre - Henderson Hospital, Hamilton, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - Ottawa Civic Hospital, Ottawa, Ontario
  - Sunnybrook and Women's College Health Science Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - University Health Network - Toronto Western Hospital, Toronto, Ontario
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - Hopital Maisonneuve Rosemont, Montreal, Quebec
  - Hopital Sacre Couer, Montreal, Quebec

REFERENCES:
- [Derived] Cook D, Sinuff T, Zytaruk N, Rabbat C, Lee A, O'Donnell M, Thabane L, Linkins L, Treleaven D, Patel R, Meade M, Crowther M, Marshall JC, Douketis J; DIRECT Investigators and Canadian Critical Care Trials Group. Event adjudication and data monitoring in an intensive care unit observational study of thromboprophylaxis. J Crit Care. 2009 Jun;24(2):168-75. doi: 10.1016/j.jcrc.2009.01.010. Epub 2009 Mar 27. PMID 19327956
- [Derived] Douketis J, Cook D, Meade M, Guyatt G, Geerts W, Skrobik Y, Albert M, Granton J, Hebert P, Pagliarello G, Marshall J, Fowler R, Freitag A, Rabbat C, Anderson D, Zytaruk N, Heels-Ansdell D, Crowther M; Canadian Critical Care Trials Group. Prophylaxis against deep vein thrombosis in critically ill patients with severe renal insufficiency with the low-molecular-weight heparin dalteparin: an assessment of safety and pharmacodynamics: the DIRECT study. Arch Intern Med. 2008 Sep 8;168(16):1805-12. doi: 10.1001/archinte.168.16.1805. PMID 18779469
- [Derived] Cook D, Douketis J, Meade M, Guyatt G, Zytaruk N, Granton J, Skrobik Y, Albert M, Fowler R, Hebert P, Pagliarello G, Friedrich J, Freitag A, Karachi T, Rabbat C, Heels-Ansdell D, Geerts W, Crowther M; Canadian Critical Care Trials Group. Venous thromboembolism and bleeding in critically ill patients with severe renal insufficiency receiving dalteparin thromboprophylaxis: prevalence, incidence and risk factors. Crit Care. 2008;12(2):R32. doi: 10.1186/cc6810. Epub 2008 Mar 3. PMID 18315876